CLINICAL TRIAL: NCT00158366
Title: A Clinical Trial Of Weight Reduction in Schizophrenia
Brief Title: Reducing the Weight of Overweight Schizophrenia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rohan Ganguli, Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH066068 (NIH); R01MH066068 (NIH); DSIR 83-ATAP; NCT00177905 (obsolete NCT alias)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia; Obesity
Keywords: Weight Loss
MeSH Terms: conditions — Schizophrenia; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Phase 1 participants who will receive behavioral training for 14 weeks
  Interventions: Behavioral: Behavioral training
- 2 (Active Comparator): Phase 1 participants who will receive social skills training for 14 weeks
  Interventions: Behavioral: Social skills training
- 3 (Experimental): Participants in the Phase 1 behavioral training group who have a 4% or more weight loss and will be enrolled in weekly behavioral training alone for 24 months in Phase 2
  Interventions: Behavioral: Behavioral training
- 4 (Experimental): Participants in the Phase 1 behavioral training group who have a 4% or more weight loss and will be enrolled in weekly behavioral training plus biweekly booster treatments for 24 months in Phase 2
  Interventions: Behavioral: Behavioral training booster sessions

INTERVENTIONS:
Behavioral: Behavioral training — The behavioral training will teach participants ways to control their diet and increase their physical activity.
  Arms: 1; 3
Behavioral: Social skills training — The social skills training will teach participants how to indirectly control their weight by making social contacts and seeking social support.
  Arms: 2
Behavioral: Behavioral training booster sessions — During biweekly booster treatment sessions, participants will discuss their response to different diet and exercise regimens, and researchers will discuss strategies for increasing one's success with the regimens.
  Arms: 4

SUMMARY:
This study will determine the effectiveness of a group-based behavioral program for weight reduction in overweight and obese schizophrenia patients.

DETAILED DESCRIPTION:
Researchers have found a link between schizophrenia, high blood pressure, and insulin resistance; this link puts people with schizophrenia at an increased risk for diabetes and obesity. Weight reduction and maintenance is essential for decreasing these risks. Although data indicate that nonpharmacological interventions for weight loss are viable options, studies to determine their effectiveness have not been conducted. This study will determine the effectiveness of behavioral training for reducing weight in schizophrenia patients. This study will also determine the effects of weight reduction on cardiovascular risk factors in this population.

This study comprises two phases. In Phase 1, participants will be randomly assigned to receive either behavioral training or social skills training for 14 weeks. The behavioral training will teach participants ways to control their diet and increase their physical activity. The social skills training will teach participants how to indirectly control their weight by making social contacts and seeking social support. After 14 weeks, participants in the social skills training group and any participants who have not lost a specified amount of weight will complete the study; participants in the behavioral training group who have a 4% or more weight loss will be enrolled in Phase 2, a 24-month program designed to help participants maintain their weight loss. All participants in Phase 2 will continue to receive weekly behavioral training, but they will be randomly assigned to receive either behavioral training alone or behavioral training combined with biweekly booster treatments where participants discuss their response to different diet and exercise regimens and researchers discuss strategies for increasing one's success with the regimens. Interviews, self-report scales, and blood tests will be used to assess participants at study entry, after Phase 1, and at the end of the study. Assessments will include quality of life, self esteem, exercise frequency, blood pressure, serum lipids, and blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* Body mass index (BMI) greater than 27
* Stable on antipsychotic drug regimen for at least 1 month prior to study entry
* Parent or guardian willing to provide informed consent, if applicable
* Positive and negative syndrome scale score less than 90
* Willing to use acceptable methods of contraception during the study

Exclusion Criteria:

* Medical contraindication for participating in a weight reduction/exercise program
* Mental retardation
* Current enrollment in another weight management program
* Current use of weight reduction medication
* Unstable cardiovascular or thyroid disease
* Active or end-stage renal disease
* Psychiatric hospitalization within 1 month prior to study entry
* Current use of more than one anti-psychotic medication
* Pregnancy or breastfeeding

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 261 (Actual)
Dates: Start 2004-05; Primary Completion 2010-05 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Weight reduction | Measured at Week 14 and Month 24

SECONDARY OUTCOMES:
Weight maintenance | Measured at Week 14 and Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Ganguli, MD, Principal Investigator — Western Psychiatric Institute and Clinic of University of Pennsylvania Medical Center
Locations (1):
- Western Psychiatric Institute and Clinic of University of Pennsylvania Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Brar JS, Ganguli R, Pandina G, Turkoz I, Berry S, Mahmoud R. Effects of behavioral therapy on weight loss in overweight and obese patients with schizophrenia or schizoaffective disorder. J Clin Psychiatry. 2005 Feb;66(2):205-12. doi: 10.4088/jcp.v66n0208. PMID 15705006
- [Background] Ganguli R, Brar JS, Ayrton Z. Weight gain over 4 months in schizophrenia patients: a comparison of olanzapine and risperidone. Schizophr Res. 2001 Apr 30;49(3):261-7. doi: 10.1016/s0920-9964(00)00080-3. PMID 11356587
- [Background] Ganguli R. Weight gain associated with antipsychotic drugs. J Clin Psychiatry. 1999;60 Suppl 21:20-4. PMID 10548138
- [Derived] Janney CA, Ganguli R, Richardson CR, Holleman RG, Tang G, Cauley JA, Kriska AM. Sedentary behavior and psychiatric symptoms in overweight and obese adults with schizophrenia and schizoaffective disorders (WAIST Study). Schizophr Res. 2013 Apr;145(1-3):63-8. doi: 10.1016/j.schres.2013.01.010. Epub 2013 Feb 12. PMID 23410710